CLINICAL TRIAL: NCT05152498
Title: Forming a Comprehensive Treatment Plan for the Treatment of Hepatitis B Virus Related Hepatocellular Carcinoma With the Core Principles of Fuzheng Jiedu Huayu
Brief Title: Fu Zheng Jie Du Hua Yu Principle For Treatment Of Severe HBV Related Hepatocellular Carcinoma (FZJDHYPFTOSHBVHCC)
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Zhiyun Yang, Archiater, Professor, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BeijingDH-YZY
Record Dates: First submitted 2021-12-08; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fu Zheng Jie Du Hua Yu therapy (Experimental)
  Interventions: Drug: Fu Zheng Jie Du Hua Yu therapy
- Routine medical care (Experimental)
  Interventions: Drug: Fu Zheng Jie Du Hua Yu therapy

INTERVENTIONS:
Drug: Fu Zheng Jie Du Hua Yu therapy — Fu Zheng Jie Du Hua Yu is a Chinese herbal compound

SUMMARY:
The treatment of HBV related hepatocellular carcinoma has always been a worldwide problem. The aim of this study is to alleviate the progression of hepatitis B related hepatocellular carcinoma by the Chinese medicine "Fu Zheng Jie Du Hua Yu" Principle.

ELIGIBILITY:
Inclusion Criteria:

* Meet the criteria of hepatocellular carcinoma
* Ages Eligible for Study: ≤75 years old;
* Informed consent from the patient.

Exclusion Criteria:

* Serious problem of heart, lung, or kidney with severe dysfunction;
* Pregnant or child breast feeding women;
* Mental or cognitive disorders;
* Participating in other drug trials;
* Who are allergic to the study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to Progression | 1 year

SECONDARY OUTCOMES:
overall survival | 1 year
progression-free survival | 1 year
complete response | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiyun Yang, Beijing, Beijing Municipality, China